CLINICAL TRIAL: NCT03824054
Title: Evaluation of Quality of Life and Gastrointestinal Well-being in Patients Undergoing Colorectal Resection for Deep Infiltrating Endometriosis. Retrospective Observational Cohort Study
Brief Title: Quality of Life in Patients Undergoing Colorectal Resection for Deep Infiltrating Endometriosis
Acronym: ENDO-RESECT
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Other Study IDs: CICOG-31-10-18\100
Record Dates: First submitted 2018-12-02; First posted 2019-01-31 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Endometriosis
Keywords: deep infiltrating endometriosis; colorectal resection; quality of life
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal resection arm: Patients affected by symptomatic deep infiltrating endometriosis involving the bowel and submitted to colo-rectal resection
  Interventions: Procedure: colorectal resection

INTERVENTIONS:
Procedure: colorectal resection — Surgery includes laparoscopic resection of all visible endometriosis, including resection of the affected bowel with primary anastomosis
  Other Names: ileostomy creation

SUMMARY:
The aim of this study is to evaluate the quality of life of patients undergoing colorectal resection for deep infiltrating endometriosis of the bowel. Questionnaires about pre operative status have been submitted retrospectively, while post operative questionnaires have been submitted prospectively during last follow up visit

DETAILED DESCRIPTION:
All patients fit for the study will be asked to complete a visual analogue scales (VAS) for dysmenorrhea, deep dyspaurenia, dysuria, dyschesia and chronic pelvic pain (CPP) Patients will fill in the Endometriosis QoL Questionnaire (EHP30), the gastrointestinal well-being questionnaires Bristol Stool Chart, GSCG (Gastrointestinal Symptom Rating Scale), STAY (1 and 2), the Psychological General Well-Being Index (PGWBI), Generalized Self-Efficacy, CD-RISC - Connor-Davidson scale about their pre operative and actual status.

Surgery includes laparoscopic resection of all visible endometriosis, including resection of the affected bowel with primary anastomosis Perioperative and post-operative complications will be collected using the Extended Clavien-Dindo classification of surgical complications divided in early (within 30 days after surgery onset) and late (over 30 days after surgery onset).

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years
* Clinical diagnosis of deep endometriosis infiltrating the bowel
* Women undergoing surgical removal with colorectal resection with or without loop ileostomy creation

Exclusion Criteria:

* History of previous or ongoing neoplastic pathology
* Contraindications to surgical intervention
* Not complete eradicating surgery
* Psychiatric disorders
* Surgical, spontaneous or pharmacological menopause - Intestinal surgery different from segmental bowel resection and colorectal anastomosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients affected by symptomatic deep infiltrating endometriosis involving the bowel and candidate to colo-rectal resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-10-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Pre-post colorectal resection-and-anastomosis evaluation of gastrointestinal symptoms (stipsi, dyschezia, regurgitation, nausea and vomit, abdominal distension and belching) | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal-resection-and-anastomosis evaluation (mean difference or percentage variation) of stipsi, dyschezia, regurgitation, nausea and vomit, abdominal distension and belching, through the administration of the GSRS (Gastrointestinal Symptom Rating Scale) to patients. The GSRS is a disease-specific instrument that includes 15 items combined into five-symptom clusters addressing different gastrointestinal symptoms. The five-symptom clusters depict reflux, abdominal pain, indigestion, diarrhoea and constipation. The GSRS has a seven-graded scale where 1 represents absence of bothersome symptoms and 7 represents very bothersome symptoms

SECONDARY OUTCOMES:
Pre-post colorectal resection-and-anastomosis evaluation of anxiety, depression, positivity and well-being, self control, general health and vitality | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal-resection-and-anastomosis evaluation (mean difference or percentage variation) of anxiety, depression, positivity and well-being, self control, general health and vitality, through the administration of the PGWBI (Psychological General Well-Being Index) to patients. The PGWBI is a brief self-administered questionnaire which contains 20 items rated on a six-point scale, where a higher score indicates a better quality of life and measures six mood states (anxiety, depressed mood, positive well-being, self-control, general health, vitality). The six mood states are scored as follows: 25 for anxiety, 20 for positive well-being and vitality and 15 for remaining
Pre-post colorectal resection-and-anastomosis evaluation of the coping ability of daily living | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal-resection-and-anastomosis evaluation (mean difference or percentage variation) of the coping ability of daily living, through the administration of the GSE (General Self-Efficacy Scale) to patients.
  The GSE consists of 10 items, with a 4-point Likert scale ranging from 1 (I Completely Disagree) to 4 (I Completely Agree), aimed at identifying, as expressed in the introduction, self-efficacy beliefs in view of difficult situations
Pre-post colorectal-resection-and-anastomosis evaluation of patients ability to "thrive in the face of adversity" | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal-resection-and-anastomosis evaluation (mean difference or percentage variation) of the ability to "thrive in the face of adversity", through the administration of the CD-RISC (Connor-Davidson Resilience Scale) to patients.
  The CD-RISC contains 25 items, all of which carry a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The scale is rated based on how the subject has felt over the past month. The total score ranges from 0-100, with higher scores reflecting greater resilience
Pre-post colorectal resection-and-anastomosis evaluation of the effects that endometriosis can have on women's lives (includes work and family life, sexual life, fertility issues) | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal resection-and-anastomosis evaluation of the effects that endometriosis can have on women's lives (work and family life, sexual life, fertility issues), through the administration of the EHP-30(Endometriosis Health Profile questionnaire).The EHP-30 consists of a 30-item core questionnaire, covers five subscales (11 items on pain, 6 on control and powerlessness, 6 on emotions, 4 on social support, 3 on self-image), and a second 23-item modular questionnaire contains six subscales (5 items on work life, 2 on relationship with children, 5 on sexual intercourse, 4 on medical profession, 3 on treatment and 4 on infertility). Response categories are rated on a five-point Likert scale (0-4), and items within each subscale are summed to create a raw-score.Each raw scale is translated into a score ranging from 0(best possible health status) to 100 by dividing the total raw scores in each subscale by the maximum possible raw-score within the subscale and multiplying it by 100
Pre-post colorectal-resection-and-anastomosis evaluation of the menstrual pain | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Pre-post colorectal-resection-and-anastomosis evaluation (mean difference or percentage variation) of the menstrual pain, through the administration of the VAS (Visual Analogic Scale) to patients. The VAS using a 10-cm line represented the continuum of the patient's opinion of the degree of pain. One extremity of the line represented "unbearable pain," and the other extremity represented "no pain at all." The participants were asked to rate the degree of pain by making a mark on the line. The scores received from the scale were classified into mild dysmenorrhea if it was between 1 and 3 points moderate between 4 and 7 points, and severe between 8 and 10 points
Prevalence of post-operative complications (rectovaginal fistulae, bowel leakage, pelvic abscesses, and postoperative bleeding) | from surgery to last follow up visit (which varies from 12 months to a maximum of 157 months)
  Perioperative and post-operative complications were collected using the Extended Clavien-Dindo classification of surgical complications divided in early (within 30 days after surgery onset) and late (over 30 days after surgery onset). Major complications were defined as those requiring surgical, endoscopic, or radiological intervention (grade III or higher according to the Clavien-Dindo classification), and include rectovaginal fistulae, bowel leakage, pelvic abscesses, and postoperative bleeding after surgery. Minor complications were defined as those that could be solved with a conservative approach (Clavien-Dindo grade I and II)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cosentino, MD, Principal Investigator — francesco.cosentino@fgps.it
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turco LC, Scaldaferri F, Chiantera V, Cianci S, Ercoli A, Fagotti A, Fanfani F, Ferrandina G, Nicolotti N, Tamburrano A, Vargiu V, Scambia G, Cosentino F. Long-term evaluation of quality of life and gastrointestinal well-being after segmental colo-rectal resection for deep infiltrating endometriosis (ENDO-RESECT QoL). Arch Gynecol Obstet. 2020 Jan;301(1):217-228. doi: 10.1007/s00404-019-05382-8. Epub 2019 Nov 22. PMID 31758304